CLINICAL TRIAL: NCT02276053
Title: A Noninterventional Study of Vimpat® (Lacosamide) as Adjunctive Antiepileptic Drug Therapy in Patients With Brain Tumor-related Epilepsy
Brief Title: Study of Lacosamide as an Adjunctive Drug Treatment for Epilepsy in Patients With Brain Tumors
Acronym: VIBES
Status: Completed | Type: Observational
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: EP0045
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Brain Tumor Related Epilepsy (BTRE)
Keywords: Epilepsy; Brain tumor; lacosamide (LCM); Anti-Epileptic Drugs (AEDs)
MeSH Terms: conditions — Epilepsy; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BTRE patients: Patients with brain tumor-related epilepsy (BTRE) routinely treated with lacosamide as add on to one or two baseline anti-epileptic drugs.

SUMMARY:
This study is being conducted to find out whether lacosamide (a drug to treat epilepsy) is effective in routine clinical practice for patients with epilepsy caused by a brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patient has never been treated with lacosamide (LCM) prior to this non-interventional study (NIS) or treatment with LCM for the first time started no earlier than 7 days prior to enrollment in this NIS
* The decision by the treating physician to prescribe LCM falls within current standard clinical practice, and the treatment decision is clearly separated from the decision to consider inclusion of the patient in the NIS
* A Patient Data Consent form is signed and dated by the patient and/or by the parent(s) or legal representative
* Patient is a male or female ≥ 16 years of age
* Patient must have a diagnosis of brain tumor-related epilepsy (BTRE) secondary to low-grade glioma (World Health Organization Grade 1 to 2 at time of enrollment)
* Patient has a retrospective Baseline seizure frequency of at least 1 partial-onset seizure in the 8 weeks prior to Visit 1 (enrollment/ Baseline visit)
* Patient does not have a previous diagnosis of epilepsy before tumor onset
* Patient does not have brain metastases
* Patient has a Karnofsky performance status scale index ≥ 60 %
* Patient is currently taking only 1-2 Baseline anti-epileptic drugs (AEDs) for epilepsy, other than LCM
* Patient has received a maximum of 4 different lifetime AEDs ever before entering the NIS

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 16 years of age with brain tumor related epilepsy secondary to low grade tumor starting with lacosamide as add-on to one or two baseline anti-epileptic drugs.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-11-27 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (24):
- France (3):
  - 337, Lille
  - 334, Lyon
  - 335, Paris
- Germany (4):
  - 491, Bonn
  - 493, Freiburg im Breisgau
  - 492, Regensburg
  - 494, Tübingen
- Italy (9):
  - 398, Ancona
  - 397, Lecco
  - 394, Milan
  - 391, Perugia
  - 392, Roma
  - 396, Roma
  - 395, San Fermo della Battaglia
  - 393, Torino
  - 399, Venezia
- Netherlands (3):
  - 311, Amsterdam
  - 312, Leidschendam
  - 314, Tilburg
- Spain (2):
  - 341, Badalona
  - 344, Barcelona
- United Kingdom (3):
  - 443, Edgbaston
  - 441, Edinburgh
  - 442, London

REFERENCES:
- [Background] Ruda R, Houillier C, Maschio M, Reijneveld JC, Hellot S, De Backer M, Chan J, Joeres L, Leunikava I, Glas M, Grant R. Effectiveness and tolerability of lacosamide as add-on therapy in patients with brain tumor-related epilepsy: Results from a prospective, noninterventional study in European clinical practice (VIBES). Epilepsia. 2020 Apr;61(4):647-656. doi: 10.1111/epi.16486. PMID 32329527
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in November 2014 and concluded in December 2017.
Pre-assignment Details: The Participant Flow refers to the Safety Set (SS), which was defined as all patients included in the study receiving treatment with LCM at least once in the study.
Groups:
- Lacosamide: Patients with brain tumor-related epilepsy (BTRE), secondary to low-grade glioma (WHO Grade 1 to 2) and with at least 1 partial-onset seizure in the 8 weeks prior to start of lacosamide (LCM) treatment, routinely treated with lacosamide as add on to one or two baseline anti-epileptic drugs (AEDs) and who were included in the Safety Set (SS).
Period: Overall Study
Arm/Group | Lacosamide
Started | 93
Completed | 79
Not Completed | 14
Not completed — Death | 2
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patient does not meet selection criteria | 3
Not completed — Patient needs to increase baseline AED | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Safety Set (SS), which was defined as all patients included in the study receiving treatment with LCM at least once in the study.
Arm/Group | Lacosamide
Number analyzed (Participants) | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 82
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Response at the End of the 6-month Observation Period
Description: A responder is a patient experiencing a 50 % or greater reduction in partial onset seizure frequency from Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all patients in the Safety Set (SS) who had at least 1 post Baseline Patient Global Impression of Change (PGIC) or seizure assessment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Lacosamide (FAS): Patients with BTRE, secondary to low-grade glioma (WHO Grade 1 to 2) and with at least 1 partial-onset seizure in the 8 weeks prior to start of LCM treatment, routinely treated with lacosamide as add on to one or two baseline AEDs and who were included in the Full Analysis Set (FAS), having at least one post-Baseline Patient Global Impression of Change or seizure assessment.
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 86
percentage of patients | 76.7 [66.4 to 85.2]

2. Primary Outcome: Patient Global Impression of Change (PGIC) Rating at Visit 3
Description: The Patient Global Impression of Change scale is a seven-point scale for patients to rate their general health status at the end of the study compared to how they felt before entering the study. Scores 1 to 3 mean improvement, score 4 means no change, and scores 5 to 7 mean worsening.
  The category 'Improved' represents the sum of Very Much Improved, Much Improved, and Minimally Improved.
  The category 'Worsened' represents the sum of Minimally Worse, Much Worse, and Very Much Worse.
Time Frame: Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 76
Participants
  Improved | 49
  No change | 17
  Worsened | 10

3. Secondary Outcome: Percentage of Patients With Retention on Lacosamide (LCM) at the End of the 6-month Observation Period
Description: The retention rate was defined as the percentage of patients remaining in the study and on Lacosamide treatment for 6 months (6 month retention rate).
Time Frame: Visit 3 (Month 6 or end of Observation Period)
Population: The analysis was performed on the Safety Set (SS), which included all patients who received treatment with lacosamide (LCM) at least once in the study.
Measure: Number; unit: percentage of patients
Groups:
- Lacosamide (SS): Patients with BTRE, secondary to low-grade glioma (WHO Grade 1 to 2) and with at least 1 partial-onset seizure in the 8 weeks prior to start of LCM treatment, routinely treated with lacosamide as add on to one or two baseline AEDs and who were included in the SS.
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 93
percentage of patients | 63.4
Statistical Analysis 1: Comparison: Lacosamide (SS); The retention rate was derived using Kaplan-Meier methodology where patients who completed the study were censored at the date of last administration of LCM in the study; Test type: Other; Retention rate = 86.0, 95% CI 2-sided [79.0 to 93.1] — Confidence intervals for the 6-month retention rate were calculated using Greenwood's formula. Addition of a note: Not all patients had an Observation Period of 6 months

4. Secondary Outcome: Time to Discontinuation of Lacosamide (LCM) Treatment From the Date of First Dose of LCM
Description: Time between first dose of LCM to discontinuation of LCM treatment was measured in days.
Time Frame: From first dose to discontinuation, over a 6-month Observation Period
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 93
days | NA [NA to NA] — Due to low number of participants with events, Kaplan-Meier estimation of percentage of event-free subjects was high and corresponding standard error was small, preventing estimation of median time to event and 95% confidence interval boundaries.

5. Secondary Outcome: Change From Visit 1 (Baseline) to Visit 3 (Month 6 or End of Observation Period) in the 5 Level EuroQol-5 Dimension Quality of Life Assessment (EQ-5D-5L) Visual Analogue Scale (VAS) Score
Description: EQ-5D-5L: 5 Level EuroQol-5 Dimension Quality of Life Assessment is a patient-completed questionnaire for patients to rate their quality of life status in five questions and a 0 (no pain) - 100 (worst pain) score vertical visual analogue scale. The Change from Baseline is calculated for this endpoint, negative values indicate improvement and positive values indicate worsening.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 72
scores on a scale | 1.3 (16.4)

6. Secondary Outcome: Change From Visit 1 (Baseline) to Visit 3 (Month 6 or End of Observation Period) in the 5 Level EuroQol-5 Dimension Quality of Life Assessment (EQ-5D-5L) Change in Utility as Converted From the 5 Dimensions
Description: EQ-5D-5L: 5 Level EuroQol-5 descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression with five response levels for each dimension: no problems, slight problems, moderate problems, severe problems and extreme problems. This 5-dimension health status is converted into a numerical utility value using the UK value set, as per EuroQOL guidelines. The utility score ranges from 0 to 1 (0=worst imaginable health state, 1=best imaginable health state). The Change from Baseline is calculated for this endpoint, negative values indicate worsening and positive values indicate improvement.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 73
scores on a scale | -0.01 (0.20)

7. Secondary Outcome: Change From Visit 1 (Baseline) to Visit 3 (Month 6 or End of Observation Period) in the M.D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT)
Description: MDASI-BT is a 2-part patient completed questionnaire where patients have to answer 22 questions about their brain tumor-related symptoms and 6 questions about how these symptoms interfere with their life. The mean core symptom severity is derived as the mean of the 13 core symptom items, the mean module symptom severity is derived as the mean of the 9 brain tumor specific symptom items and the mean total symptom severity is derived as the mean of all 22 symptom items. The mean interference is derived as the mean of the 6 interference items. For each score, at least 50% of the items needs to be answered for the score to be calculated. Mean core, mean module and mean total symptom severity scores are ranging from 0 to 10 (0=not present 10=as bad as you can imagine). Mean interference score is ranging from 0 to 10 (0= did not interfere 10= interfered completely). The Change from Baseline is calculated, negative values indicate improvement, positive values indicate worsening.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 73
scores on a scale
  Mean core symptom severity | 0.1 (1.3)
  Mean module symptom severity: number analyzed (Participants) | 70
  Mean module symptom severity | -0.1 (1.6)
  Mean total severity | 0.0 (1.2)
  Mean interference: number analyzed (Participants) | 70
  Mean interference | -0.5 (2.4)

8. Secondary Outcome: Actual Change From Visit 1 (Baseline) to Visit 3 (Month 6 or End of Observation Period) in Seizure Frequency (Seizures Per 28 Days)
Description: The actual change in seizure frequency from Baseline to Month 6 is calculated as the seizure frequency at Month 6 minus the seizure frequence at Baseline.
  The seizure frequency at each time point is calculated as number of seizures per 28 days.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seizures per 28 days
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 78
seizures per 28 days | -2.9 [-9.1 to -0.9]

9. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency
Description: The percentage change from Baseline to Month 6 in seizure frequency is the actual change in seizure frequency for this period compared to the Baseline seizure frequency, which is considered 100 %.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 78
percent change | -85.2 [-100.0 to -55.5]

10. Secondary Outcome: Percentage of Patients With Seizure-free Status (Yes/No) at the End of the 6-month Observational Period
Description: Percentage of patients achieving a seizure-free status at the end of the 6-month Observation Period.
Time Frame: Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 86
percentage of patients | 34.9 [24.9 to 45.9]

11. Secondary Outcome: Discontinuation Rate of Lacosamide (LCM) Due to Adverse Drug Reactions (ADRs)
Description: Discontinuation rate due to ADRs is the number of patients that discontinued from the study and from LCM treatment due to ADRs during the 6 months of observation.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 93
Participants | 5

12. Secondary Outcome: Discontinuation Rate of Lacosamide (LCM) Due to Lack of Effectiveness
Description: Discontinuation rate due to lack of effectiveness is the number of patients that discontinued from the study and from LCM treatment due to lack of effectiveness during the 6 months of observation.
Time Frame: Visit 1 (Baseline) to Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 93
Participants | 7

13. Secondary Outcome: Clinical Global Impression of Change (CGIC) Rating at Visit 3 (Month 6 or End of Observation Period)
Description: The Clinical Global Impression of Change is a seven-point scale for the treating physician to rate the patient's general health status at the end of the study compared to how the patient felt before entering the study. Scores 1 to 3 mean improvement, score 4 means no change, and scores 5 to 7 mean worsening.
  The category 'Improved' represents the sum of Very Much Improved, Much Improved, and Minimally Improved.
  The category 'Worsened' represents the sum of Minimally Worse, Much Worse, and Very Much Worse.
Time Frame: Visit 3 (Month 6 or end of Observation Period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 81
Participants
  Impoved | 52
  No change | 19
  Worsened | 10

ADVERSE EVENTS:
Time Frame: From Baseline and up to month 6
Arm/Group | Lacosamide (SS)
All-Cause Mortality (participants affected / at risk) | 2/93
Serious Adverse Events (participants affected / at risk) | 5/93
Other Adverse Events (participants affected / at risk) | 9/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=93)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=93)
Vertigo (Ear and labyrinth disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT02276053/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT02276053/SAP_001.pdf